CLINICAL TRIAL: NCT04411186
Title: A Trial of Adding Lung Protective Strategies to Existing Enhanced Recovery After Surgery (ERAS) Protocols and Its Effects on Improving Post-Operative Lung Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, David Gutman, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00094011
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Surgery; Hepatobiliary Surgery
MeSH Terms: interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Enhanced Recovery After Surgery (ERAS) Protocol (Active Comparator): Control for this study will be the standard MUSC ERAS protocol - fluid intake, hydration, anti-emetics, pain control, and several other considerations.
  Interventions: Procedure: Standard Enhanced Recovery After Surgery (ERAS) Protocol
- ERAS and 5 Lung Protective Interventions (Experimental): The standard MUSC ERAS protocol - fluid intake, hydration, anti-emetics, pain control, and several other considerations. The subject will also receive the following lung protective interventions:
  1. Pressure control ventilation-volume guaranteed (PCV-VG) ventilation at approximately 7cc/kg of predicted body weight (derived from combination of sex and height)
  2. Positive end-expiratory pressure (PEEP) 7cm H2O5
  3. Immediately post intubation recruitment breath (30cm water for 30 seconds)
  4. Every 1 hour recruitment breath (30cm water for 30 seconds)
  5. 40% FIO2 initially - titrate up as necessary to maintain SPO2 >94%
  Interventions: Procedure: ERAS and 5 Lung Protective Interventions

INTERVENTIONS:
Procedure: Standard Enhanced Recovery After Surgery (ERAS) Protocol — Subjects receive standard MUSC ERAS protocol - fluid intake, hydration, anti-emetics, pain control, and several other considerations.
  Arms: Standard Enhanced Recovery After Surgery (ERAS) Protocol
Procedure: ERAS and 5 Lung Protective Interventions — Subjects will receive the standard MUSC ERAS protocol - fluid intake, hydration, anti-emetics, pain control, and several other considerations. The subject will also receive the following lung protective interventions:
  Pressure control ventilation-volume guaranteed (PCV-VG) ventilation at approximately 7cc/kg of predicted body weight (derived from combination of sex and height) Positive end-expiratory pressure (PEEP) 7cm H2O5 Immediately post intubation recruitment breath (30cm water for 30 seconds) Every 1 hour recruitment breath (30cm water for 30 seconds) 40% FIO2 initially - titrate up as necessary to maintain SPO2 >94%
  Arms: ERAS and 5 Lung Protective Interventions

SUMMARY:
The objective of this study is to determine whether the addition of lung protective strategies to existing enhanced recovery after surgery (ERAS) protocols for colorectal surgeries and hepatobiliary surgeries will improve post-operative lung function.

ELIGIBILITY:
Inclusion Criteria:

* All subjects going for scheduled colorectal or hepatobiliary surgery at the MUSC ART hospital who would normally be utilizing the existing ERAS protocols
* English speaking
* Able to give informed consent
* Ages 18 years and older

Exclusion Criteria:

* Emergency cases
* Pregnant subjects-confirmed by pre-operative urine pregnancy test
* Subjects with unique lung pathologies including, but not limited to: advanced pulmonary fibrosis, lung transplantation recipients, end stage COPD, pulmonary Hypertension
* Subjects on home O2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gutman, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ERAS and 5 Lung Protective Interventions: The standard MUSC ERAS protocol - fluid intake, hydration, anti-emetics, pain control, and several other considerations. The subject will also receive the following lung protective interventions:
  1. Pressure control ventilation-volume guaranteed (PCV-VG) ventilation at approximately 7cc/kg of predicted body weight (derived from combination of sex and height)
  2. Positive end-expiratory pressure (PEEP) 7cm H2O5
  3. Immediately post intubation recruitment breath (30cm water for 30 seconds)
  4. Every 1 hour recruitment breath (30cm water for 30 seconds)
  5. 40% FIO2 initially - titrate up as necessary to maintain SPO2 >94%
  ERAS and 5 Lung Protective Interventions: Subjects will receive the standard MUSC ERAS protocol - fluid intake, hydration, anti-emetics, pain control, and several other considerations. The subject will also receive the following lung protective interventions:
  Pressure control ventilation-volume guaranteed (PCV-VG) ventilation at approximately 7cc/kg of predicted body weight (derived from combination of sex and height) Positive end-expiratory pressure (PEEP) 7cm H2O5 Immediately post intubation recruitment breath (30cm water for 30 seconds) Every 1 hour recruitment breath (30cm water for 30 seconds) 40% FIO2 initially - titrate up as necessary to maintain SPO2 >94%
Period: Overall Study
Arm/Group | Standard Enhanced Recovery After Surgery (ERAS) Protocol | ERAS and 5 Lung Protective Interventions
Started | 50 | 50
Completed | 50 | 49 (one patient was withdrawn)
Not Completed | 0 | 1
Not completed — Withdrawn due to protocol violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Enhanced Recovery After Surgery (ERAS) Protocol | ERAS and 5 Lung Protective Interventions | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Customized [Count of Participants; unit: Participants]
  ≤ 30 years | 2 | 1 | 3
  31-50 years | 9 | 9 | 18
  51-70 years | 28 | 26 | 54
  ≥ 71 years | 11 | 13 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 27 | 19 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 49 | 99
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 42 | 40 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  Underweight (<18.5) | 2 | 3 | 5
  Normal ((≥ 18.5, < 25) | 14 | 15 | 29
  Overweight (≥ 25, < 30) | 19 | 17 | 36
  Obese (≥ 30) | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Capacity
Description: The primary outcome of interest is the inspiratory capacity obtained in the PACU via the incentive spirometer.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Standard Enhanced Recovery After Surgery (ERAS) Protocol | ERAS and 5 Lung Protective Interventions
Number analyzed (Participants) | 50 | 49
mL
  Preoperative incentive spirometry (average) | 2,043.3 (628.4) | 2,012.2 (895.2)
  Postoperative incentive spirometry 30 min (average) | 1,195.2 (715.0) | 1,233.3 (894.1)
  Postoperative incentive spirometry 1 h (average) | 1,313.9 (618.1) | 1,387.3 (975.3)
  Postoperative incentive spirometry 2 h (average) | 1,376.3 (651.2) | 1,454.8 (906.4)
  Postoperative incentive spirometry total (average) | 1,253.5 (593.7) | 1,390.4 (964.9)

2. Secondary Outcome: Oxygen Saturation (SPO2) Trends
Description: Numerical value for SPO2 trends in 15 min intervals in the Post Operative Care Unit (PACU)
Time Frame: 2 hours
Population: Data was for this outcome was not documented by nursing staff in the medical record, therefore this outcome was unable to be included and analyzed.
Arm/Group | Standard Enhanced Recovery After Surgery (ERAS) Protocol | ERAS and 5 Lung Protective Interventions
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Supplemental Oxygen Requirements
Description: Recording of use or lack thereof of supplemental oxygen in PACU in 15 minute intervals.
Time Frame: 2 hours
Population: as for outcome 2
Arm/Group | Standard Enhanced Recovery After Surgery (ERAS) Protocol | ERAS and 5 Lung Protective Interventions
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent and enrollment through each patient's completion of the study which was until they leave the PACU, or until two hours has passed, whichever was less.
Arm/Group | Standard Enhanced Recovery After Surgery (ERAS) Protocol | ERAS and 5 Lung Protective Interventions
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

LIMITATIONS AND CAVEATS:
Limitations to the study included difficulties with obtaining all data points during the post-anesthesia care unit (PACU) timeframe, specifically the use of supplemental oxygen in the PACU, therefore fewer conclusions can be drawn without this secondary outcome data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/86/NCT04411186/Prot_SAP_000.pdf